CLINICAL TRIAL: NCT06158022
Title: Determination of ED90s of Phenylephrine and Norepinephrine Infusion for Strict Blood Pressure Management Targets in Preeclamptic Patients Undergoing Cesarean Section: A Randomized Sequential Allocation Study
Brief Title: ED90 of Norepinephrine and Phenylephrine Infusions in Preeclamptic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Yi Chen-2024-11
Record Dates: First submitted 2023-11-25; First posted 2023-12-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Adverse Effect
MeSH Terms: interventions — Norepinephrine; Vasoconstrictor Agents; Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Norepinephrine group (Experimental): The maternal systolic blood pressure was consistently maintained above 90% of the preoperative baseline value from the initiation of spinal anesthesia until fetal delivery.
  Interventions: Drug: Norepinephrine
- Phenylephrine group (Experimental): The maternal systolic blood pressure was consistently maintained above 90% of the preoperative baseline value from the initiation of spinal anesthesia until fetal delivery.
  Interventions: Drug: Phenylephrine

INTERVENTIONS:
Drug: Norepinephrine — An initial infusion dose of prophylactic norepinephrine (0.05 ug/kg/min) simultaneous with spinal anesthesia. The dose administered to subsequent patients varied by increments or decrements of 0.01 ug/kg/min of prophylactic norepinephrine according to the responses of previous patients according to the up-down sequential allocation.
  Other Names: Vasopressor
  Arms: Norepinephrine group
Drug: Phenylephrine — An initial infusion dose of prophylactic phenylephrine (0.5 ug/kg/min) simultaneous with spinal anesthesia. The dose administered to subsequent patients varied by increments or decrements of 0.1 ug/kg/min of prophylactic phenylephrine according to the responses of previous patients according to the up-down sequential allocation.
  Other Names: Vasopressor
  Arms: Phenylephrine group

SUMMARY:
The objective of this study is to investigate the ED90 of norepinephrine and phenylephrine infusions for preventing postspinal anesthesia hypotension under intensive treatment in preeclamptic patients during cesarean section

DETAILED DESCRIPTION:
Post-spinal anesthesia hypotension is a frequent complication during spinal anesthesia for cesarean section. The incidence of post-spinal anesthesia hypotension is as high as 62.1-89.7% if prophylactic measures are not taken. The 2016 ASA guidelines for obstetric anesthesia suggest avoiding hypotension following spinal anesthesia in women and emphasize the use of vasopressors, specifically alpha-receptor agonists, as the preferred strategy to prevent and manage post-spinal anesthesia hypotension. The 2018 International Consensus in the United Kingdom and Northern Ireland recommends maintaining maternal systolic blood pressure above 90% of the baseline value following lumbar anesthesia, while avoiding dropping below 80% of the baseline value. Currently, the threshold for maintaining blood pressure above 80% of the baseline value is widely adopted as a standard; however, limited evidence supports the advantage of sustaining maternal blood pressure above 90% of the baseline value. The objective of this study is to investigate the ED90 of norepinephrine and phenylephrine infusions for preventing postspinal anesthesia hypotension under intensive treatment in preeclamptic patients during cesarean section

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years
* Primipara or multipara
* Singleton pregnancy ≥32 weeks
* American Society of Anesthesiologists physical status classification II to III
* Scheduled for cesarean section under spinal anesthesia

Exclusion Criteria:

* Baseline blood pressure ≥160 mmHg
* Body height < 150 cm
* Body weight > 100 kg or body mass index (BMI) ≥ 40 kg/m2
* Eclampsia or chronic hypertension
* Hemoglobin < 7g/dl
* Fetal distress, or known fetal developmental anomaly

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-03 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
ED50 and ED90 | 1-15 minutes after spinal anesthesia
  The doses of prophylactic norepinephrine and phenylephrine that would be effective in preventing postspinal anesthesia hypotension in 50% (effective dose, ED 50) and 90% (ED90) of patients

SECONDARY OUTCOMES:
The incidence of post-spinal anesthesia hypotension | 1-15 minutes after spinal anesthesia.
  Systolic blood pressure (SBP) < 80% of the baseline
The incidence of severe post-spinal anesthesia hypotension. | 1-15 minutes after spinal anesthesia.
  Systolic blood pressure (SBP) < 60% of the baseline.
The incidence of bradycardia. | 1-15 minutes after spinal anesthesia.
  Heart rate < 60 beats/min.
The incidence of nausea and vomiting. | 1-15 minutes after spinal anesthesia.
  Presence of nausea and vomiting in patients after spinal anesthesia
The incidence of hypertension. | 1-15 minutes after spinal anesthesia.
  Systolic blood pressure (SBP) >120% of the baseline.
pH | Immediately after delivery
  From umbilical arterial blood gases.
Base excess (BE) | Immediately after delivery
  From umbilical arterial blood gases.
Partial pressure of oxygen (PO2) | Immediately after delivery
  From umbilical arterial blood gases.
APGAR score | 1 min after fetal delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration; 0(Worst)-10(Best)
APGAR score | 5 min after fetal delivery
  A= Appearance P=Pulse G=Grimace A=Attitude R=Respiration; 0(Worst)-10(Best)

CONTACTS AND LOCATIONS:
Overall Officials: Yi Chen, M.D., Study Chair — General Hospital of Ningxia Medical University
Locations (1):
- General hospital of Ningxia University, Yinchuan, Ningxia, China

REFERENCES:
- [Derived] Ma Y, Ma R, Shi Y, Qin R, Chen Y. Determination of ED90s of Phenylephrine and Norepinephrine Infusion for Strict Blood Pressure Management Targets in Preeclamptic Patients Undergoing Cesarean Section: A Randomized Sequential Allocation Study. Drug Des Devel Ther. 2025 Nov 1;19:9751-9757. doi: 10.2147/DDDT.S545813. eCollection 2025. PMID 41200476